CLINICAL TRIAL: NCT01679028
Title: Single- and Multiple- Dose-Escalation Study to Investigate the Safety and Tolerability of T89 in Japanese Healthy Volunteers
Brief Title: Dose-Escalate Study to Investigate the Safety and Tolerability of T89 in Japanese
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tasly Pharmaceuticals, Inc. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: T89-10-JP
Record Dates: First submitted 2012-08-24; First posted 2012-09-05 (Estimated); Results first posted 2014-11-24 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
Keywords: T89 Safety in Healthy Japanese population
MeSH Terms: interventions — T89 herbal drug

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo Group A (Placebo Comparator): 150mg Placebo Single dose
  Interventions: Drug: Placebo Group A
- T89 Group A (Experimental): 150mg T89 single dose
  Interventions: Drug: T89 Group A
- Placebo Group B (Placebo Comparator): 300mg placebo single dose
  Interventions: Drug: Placebo Group B
- T89 Group B (Experimental): 300mg T89 single dose
  Interventions: Drug: T89 Group B
- Placebo Group C (Placebo Comparator): 225mg Placebo bid for 14 days
  Interventions: Drug: Placebo Group C
- T89 Group C (Experimental): 225mg T89 bid for 14 days
  Interventions: Drug: T89 Group C

INTERVENTIONS:
Drug: T89 Group A — 150mg single dose on day 1
  Other Names: Dantonic®; Salvtonic®; Compound Danshen Dripping Pills
  Arms: T89 Group A
Drug: Placebo Group A — 150mg single dose
  Arms: Placebo Group A
Drug: Placebo Group B — 300mg single dose
  Arms: Placebo Group B
Drug: T89 Group B — 300mg single dose
  Other Names: Dantonic®; Salvtonic®; Compound Danshen Dripping Pills
  Arms: T89 Group B
Drug: Placebo Group C — 225mg bid
  Arms: Placebo Group C
Drug: T89 Group C — 225mg bid
  Other Names: Dantonic®; Salvtonic®; Compound Danshen Dripping Pills
  Arms: T89 Group C

SUMMARY:
The purpose of this study is to see how safe an investigational new drug (T89) is and how well healthy Japanese subjects tolerate it when given two single doses and a multiple dose.

DETAILED DESCRIPTION:
This is a single centre, double-blind, randomized, placebo controlled, single- and multiple- dose-escalation study.

After informed consent is obtained, subjects were evaluated with a medical history questionnaire, physical examination, blood and urine collections for clinical laboratory safety tests, urine drug screen, serum pregnancy test for each women, vital signs and ECG. The subjects who fulfill the inclusion criteria but no exclusion criteria were provisionally enrolled. For participation in this trial, subjects were instructed to avoid any prescription, over-the-counter (OTC), and alternative / complementary medications or significant changes in diet without advance permission from principal investigator. The subjects were instructed to discontinue alcohol, caffeine and bromine containing beverage/food. 20 subjects were enrolled and divided into three Groups: Group A, Group B and Group C.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female volunteers aged between 20-55 years.
2. First generation of Japanese, and live in the U.S.A. less than 5 years and maintained Japanese lifestyle.
3. The body mass index between 18 and 30 kg/m2.
4. Willing to not take alcoholic beverages, and caffeine- and the bromine-containing beverages and foods (e.g., tea, coffee, chocolate, cola, etc.) for the duration of the study beginning at the screening visit.
5. ECG with no clinically significant abnormalities.
6. No clinically significant medical history.
7. Vital signs and laboratory tests with no clinically significant abnormalities.
8. Volunteers had not taken any medication that would interfere with the procedures or interpretation of study data or compromise subject safety within 4 weeks prior to the first dose, per principal investigator discretion.
9. Volunteers must understand and be willing, able and likely to comply with all study procedures and restrictions.
10. Volunteers must be able to give voluntary written informed consent.

Exclusion Criteria:

1. History of uncontrolled, clinically significant neurologic, cardiovascular, haematological, pulmonary, hepatic, renal, metabolic, GI, urologic, immunologic, endocrine or psychiatric disease.
2. Pregnant or nursing mother - Women of childbearing potential must have a negative pregnancy test, not be breast feeding and be established on a method of contraception that in the investigator's opinion is acceptable.
3. Have on-going other treatment or medicine that may interfere with T89 or administration of similar medication within 2 weeks of entering study, per principal investigator discretion.
4. Blood donor in recent 3 months.
5. Have taken part in other clinical trials involving administration of study medications in the previous 1 month before participation.
6. Excessive alcohol use (habitually consumed more than 21 units of alcohol per week or has a history of alcohol abuse as defined by DSM-IV-TR criteria (a unit of alcohol is equal to 1 ounce of hard liquor, 5 ounces of wine or 8 ounces of beer within past two years).
7. History or evidence of habitual use of tobacco or nicotine containing products within 3 months of Screening, with the exception of light smoking (up to 5 cigarettes per day or the equivalent)
8. Known hypersensitivity to any of the ingredients of T89 or other relevant drug allergy.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-08; Primary Completion 2012-10 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason GUO, M.D., Study Director — Tasly Pharmaceuticals, Inc.
Locations (1):
- California Clinical Trial Medical Group, Glendale, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Initiation Date: Auguest 1st, 2012
  Study Completion Date: October 20th, 2012
  Location: Phase I clinical Study Center:
  California Clinical Trials Medical Group 1509 Wilson Terrace Glendale, CA 91206
Groups:
- Placebo Group A: Placebo 150mg single dose
- T89 Group A: T89 150mg single dose
- Placebo Group B: Placebo 300mg single dose
- T89 Group B: T89 300mg single dose
- Placebo Group C: Placebo 225mg bid for 14 days
- T89 Group C: T89 225mg bid for 14 days
Period: Overall Study
Arm/Group | Placebo Group A | T89 Group A | Placebo Group B | T89 Group B | Placebo Group C | T89 Group C
Started | 2 | 4 | 2 | 4 | 2 | 6
Completed | 2 | 4 | 2 | 4 | 2 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Placebo Group A: 2 T89 Group A: 4 Placebo Group B: 2 T89 Group B: 4 Placebo Group C: 2 T89 Group C: 6
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Group A | T89 Group A | Placebo Group B | T89 Group B | Placebo Group C | T89 Group C | Total
Number analyzed (Participants) | 2 | 4 | 2 | 4 | 2 | 6 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (3) | 24 (2) | 24.5 (4.9) | 24 (2.2) | 47.5 (6.4) | 40.6 (9.9) | 32.5 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Male | 2 | 4 | 2 | 4 | 2 | 5 | 19
Region of Enrollment [Number; unit: participants]
  United States | 2 | 4 | 2 | 4 | 2 | 6 | 20

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Drug Events and Serious Adverse Events
Description: the Incidence of Adverse Drug Events and serious adverse events
Time Frame: 30 days (after first dosing)
Measure: Number; unit: adverse event
Groups:
- Placebo Group A: 150 mg placebo; single dose
- T89 Group A: 150mg T89; Single dose
- Placebo Group B: 300mg Placebo; single dose
- T89 Group B: 300mg T89; single dose
- Placebo Group C: 225mg bid for 10 days
- T89 Group C: T89 225mg bid for 10 days
Arm/Group | Placebo Group A | T89 Group A | Placebo Group B | T89 Group B | Placebo Group C | T89 Group C
Number analyzed (Participants) | 2 | 4 | 2 | 4 | 2 | 6
adverse event | 0 | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: 30 days after the last dose.
Groups:
- Placebo Group A: 150 mg Placebo Single dose
- T89 Group C: T89 225mf bid for 14 days
Arm/Group | Placebo Group A | T89 Group A | Placebo Group B | T89 Group B | Placebo Group C | T89 Group C
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4 | 0/2 | 0/4 | 0/2 | 0/6
Other Adverse Events (participants affected / at risk) | 0/2 | 0/4 | 0/2 | 0/4 | 0/2 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Group A (N=2) | T89 Group A (N=4) | Placebo Group B (N=2) | T89 Group B (N=4) | Placebo Group C (N=2) | T89 Group C (N=6)
Somnolence (General disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI can be co-authored with sponsor for the publication but cannot publish the result solely.